CLINICAL TRIAL: NCT03885778
Title: An Open Label, Randomized, 2-sequence, 2-period, Single-dose Cross-over Design Clinical Trial to Evaluate the Food Effect on Pharmacokinetics of BESIVO in Healthy Adult Volunteers
Brief Title: A Food Effect Study of Besifovir in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-BVCL-402
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Food Effect; Health Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-fasted dosing followed by fed dosing (Experimental): Fasted dosing of Besifovir dipivoxil followed by fed dosing; Dosing in the fasted state followed by fed dosing
  Interventions: Drug: Besifovir dipivoxil
- B-fed dosing followed by fasted dosing (Experimental): Fed dosing of Besifovir dipivoxil followed by fasted dosing; Dosing in the fed state followed by fasted dosing
  Interventions: Drug: Besifovir dipivoxil

INTERVENTIONS:
Drug: Besifovir dipivoxil — 150mg Besifovir dipivoxil, single dose, oral
  Other Names: Besivo tab

SUMMARY:
To investigate the PK characteristics and the effect of food on the PK in healthy volunteers who receive Besifovir dipivoxil in fed versus fasted condition

DETAILED DESCRIPTION:
A randomized, open-label, 2-sequence, 2-period, single-dose cross-over clinical trial to investigate the pharmacokinetics incorporating a comparison of fed/fasted pharmacokinetics of Besifovir dipivoxil in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
2. Age of 19 to 50 years and Body Mass Index [BMI] of 18.0 to 27.0 kg/m2
3. Subject with no congenital or chronic disease and no medically symptomatic findings
4. Subject must be healthy on the basis of vital signs, 12-lead ECG, physical examination and laboratory test performed at screening.

Exclusion Criteria:

1. Medical history

   * History of clinically significant of gastrointestinal system, hepatic portal system, cardiovascular system, respiratory system, endocrine system, renal-urinary system, immunologic system, musculoskeletal system, neurological, or psychiatric system, blood tumor, ophthalmology, otolaryngology disorder(as determined by the Investigator).
   * Prior history of a gastrointestinal disorder that may affect drug absorption, distribution, metabolism and elimination (e.g., Crohn's disease, ulcer or surgery, except for simple appendectomy or hernia surgery)
2. Clinical tests

   * Systolic Blood Pressure: lower than 90mmHg or higher than 140mmHg, Diastolic Blood Pressure: lower than 60mmHg or higher than 180mmHg
   * Repeated measurement of laboratory value outside the reference range that the investigator considers to be of clinical relevance

     1. Aspartate transaminase [AST] or alanine aminotransferase [ALT] > 1.5 x upper limit of normal range
     2. Total bilirubin > 1.5 x upper limit of normal range
     3. estimated glomerular filtration rate [eGFR] < 75mL/min/1.73m2 (using Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equations)
     4. Positive screening on Hepatitis B surface antigen(HBsAg), anti-Hepatitis C virus(HCV), anti-Human immunodeficiency virus(HIV) or Syphilis reagin test
   * Subjects with clinically significant abnormalities in 12-lead ECG determined by repeated measurement
3. Allergy, hypersensitivity, and drug abuse

   * History of significant hypersensitivity to Besifovir, this drug ingredient or other drug (e.g., aspirin, antibiotics)
   * History of clinically significant allergy/hypersensitivity
   * A history of drug abuse (especially, central nervous system agents such as sleeping pills, central painkillers, opiates or psychotropic drugs) or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs(amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines)
4. The contraindication of comedication drugs and diets

   * Subject who has taken drugs for drug metabolizing enzyme induction and inhibition within 1 month before the first adminstration
   * Subject who has taken other ethical the count [ETC] drugs (including prescription of herbal medicine) within the last 14 days, or over the count [OTC] drugs within the last 10 days (as determined by the Investigators)
   * Subject who has taken abnormal meals (eg. ingestion of grapefruit juice, garlic extract, broccoli, and kale) which can affect to drug absorption, distribution, metabolism, and excretion [ADME] and supplements within 7 days prior to administration of trial medication and during the trial
   * Subject who has participated in any other bioequivalence study or clinical trial and taken other investigational products within 3 months prior to the first adminstration
5. Donation and receipt of blood

   * Subject who had whole blood donation within 2 months prior to administration of trial medication
   * Subject who had component blood donation or transfusion within 1 months prior to administration of trial medication
6. Pregnant and contraception

   * Pregnant, positive of pregnancy test or breast-feeding women
   * Subjects who do not use medically acceptable contraception during the entire period of the trial

     1. Use of intrauterine device
     2. Use of intercourse contraceptive (male or female) and spermicide
     3. Vasectomy
     4. Tubectomy, canal ligation and hysterectomy
7. Other criteria

   * Use of Xanthine (eg. green tea, coffee, black tea, coke, cocoa, chocolate, energy drink, and etc.) within 3 days prior to administration of trial medication and during the trial
   * Intake of more than 30g of alcohol per day or who can't abstain from alcohol during the trial
   * Subjects who can't quit smoking during the trial
   * Subjects who are considered to be unacceptable in this study under the opinion of the investigator.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration [Cmax] of Besifovir | Up to 24 Hours after study drug administration
  The Cmax is the maximum observed plasma concentration.
Area Under the Curve [AUC] of of Besifovir | Up to 24 Hours after study drug administration
  Area under the plasma concentration versus time curve for Besifovir

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Besifovir | Up to 24 Hours after study drug administration
  Area under the plasma concentration-time curve from time zero to infinite time
Time to reach the Cmax [Tmax] of Besifovir | Up to 24 Hours after study drug administration
  Time to reach the Cmax of Besifovir
Apparent terminal half-life [t1/2] | Up to 24 Hours after study drug administration
  apparent terminal half-life of Besifovir

OTHER OUTCOMES:
Safety of Besifovir: incidence of treatment emergent adverse event [TEAE]'s, abnormalities | Up to 14 days after last study drug administration
  Safety of Besifovir administered orally will be assessed by incidence of treatment emergent adverse event [TEAE]'s, abnormalities in vital sign assessments, ECG's, clinical laboratory assessments, and physical exams

CONTACTS AND LOCATIONS:
Overall Officials: jong-Lyul GhimK, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No